CLINICAL TRIAL: NCT05124158
Title: Association of the Severity of the Clinical Picture of COVID-19 and Psychiatric Morbidity
Brief Title: COVID-19 Severity and Psychiatric Morbidity
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Collaborators: Universidad Autonoma de Coahuila (Other)
Responsible Party: Principal Investigator, Lilia Edith Luque Esparza, Principal Investigator, Instituto Mexicano del Seguro Social
Other Study IDs: R-2021-902-025
Record Dates: First submitted 2021-11-12; First posted 2021-11-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: COVID-19; Psychiatric Disorder
Keywords: COVID-19; Psychiatric morbidity
MeSH Terms: conditions — COVID-19; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a diagnosis of COVID-19: A directed psychiatric evaluation will be carried out and 1 evaluation instrument will be applied: Global Tool for the Evaluation of Mental Health in Primary Care (GMHAT / PC).
  The Global Mental Health Assessment Tool / Primary Care (GMHAT / PC) is a computerized, semi-structured clinical interview tool developed to assess and identify mental health problems. The main diagnosis derives from the use of a hierarchical model based on ICD-10. The diagnostic program takes into account the severity of symptoms (moderate to severe). It also generates alternative diagnoses and comorbidity states based on the presence of symptoms of other disorders. In addition, it includes a suicide risk assessment.

SUMMARY:
The COVID-19 pandemic represents the most serious global health threat since the Spanish influenza, with repercussions on physical and mental health. The balance between physical and mental state is essential when establishing treatment for a critically ill patient and must be taken into account by health professionals. Therefore, the investigators hypothesize that there is an association between the severity of the clinical picture of COVID-19 and psychiatric morbidity.

Objective. Associate the severity of the clinical picture of COVID-19 with psychiatric morbidity.

Material and method. Hospitalized participants in the COVID respiratory area at the General Hospital of the Zone will be included. # 51 of Gómez Palacio, Dgo. in the period from October 1, 2021 to March 31, 2022. This is an epidemiological, observational, prospective, longitudinal, analytical study. Sociodemographic, clinical and psychiatric evaluation data will be obtained using GMHAT / PC. A statistical analysis will be carried out using descriptive statistics (frequencies, measures of central tendency and dispersion) and analytical, to evaluate the association (Chi2) and to evaluate the effect of the intervening variables (binary logistic regression and multivariate regression). The data will be analyzed in the SPSS version 21 program.

DETAILED DESCRIPTION:
Subjects who meet selection criteria entered into the COVID area will be included in the period from October 1, 2021 to March 31, 2022. A non-probabilistic convenience sampling will be carried out, occluding all patients who agree to participate and meet the criteria of selection.

Patients entering the COVID area will be invited to participate in the study. Participants will be questioned about the selection criteria, and if they are eligible to be included in the study, they will be given the letter of informed consent for reading, clarification of doubts and signature. Each participant will receive a copy of the informed consent letter, this copy will remain in the COVID area until the participant is discharged. The researcher's copy will be handled under the biosafety standards established in the institute for materials and documents in contact with COVID patients.

Information about their general data and conventional medical history will be obtained through direct questioning and review of the medical record and a brief neuropsychiatric evaluation will be performed. The severity data of the COVID clinical picture and clinical evolution will be obtained from the records in the electronic medical record. The evaluation of psychiatric morbidities using the GMHAT / PC will be carried out later, prior to feeding the database.

The information obtained will be emptied into an Excel database for subsequent statistical analysis with the IBM SPSS STATISTICS program. The information of the study will remain confidential, the identity of the participants will be protected through the use of the initials of the participant's name. The data collected will be in charge of the researcher for safekeeping. The management of the information from the data collection sheets will be organized by folios.

ELIGIBILITY:
Inclusion Criteria:

* Beneficiaries in the COVID respiratory area of HGZ No.51
* COVID-19 diagnosis confirmed by PCR.
* Complete neuropsychiatric medical history data that allows the evaluation of the psychiatric status using GMHAT / PC
* Accept to participate in the study and sign the informed consent.

Exclusion Criteria:

* Pre-existing neuropsychiatric diseases and under psychiatric medical treatment.
* History of psychotropic use and / or withdrawal syndrome.
* Incomplete file data or that do not allow the assessment of the severity of the clinical picture of COVID-19 upon admission to the respiratory area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Beneficiaries admitted to the COVID respiratory area of HGZ No.51 in the period from October 01, 2021 to March 31, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Degree of severity of the clinical picture of COVID-19 | Duration of hospitalization (20 days)
  Severity of COVID-19 according to the clinical and paraclinical parameters established by the WHO (Mild, Moderate, Severe, Critical)
Number of participants with depression | Duration of hospitalization (20 days)
  According to the result of the psychiatric evaluation using GMHAT/PC: Absent or Present
Number of participants with anxiety | Evaluation at hospital admission (2 hours)
  According to the result of the psychiatric evaluation using GMHAT/PC: Absent or Present
Number of participants with panic disorder | Evaluation at hospital admission (2 hours)
  According to the result of the psychiatric evaluation using GMHAT/PC: Absent or Present
Number of participants with psychosis | Evaluation at hospital admission (2 hours)
  According to the result of the psychiatric evaluation using GMHAT/PC: Absent or Present

SECONDARY OUTCOMES:
Clinical evolution of the participants measured by clinical and paraclinical parameters | Duration of hospitalization (20 days)
  Worsening or improvement of the disease measurable by observable and diagnosable signs and symptoms according to the clinical and paraclinical parameters established by the WHO.

CONTACTS AND LOCATIONS:
Overall Officials: Lilia E Luque Esparza, Dra., Principal Investigator — IMSS
Locations (1):
- Instituto Méxicano del Seguro Social, Gómez Palacio, Durango, Mexico

IPD SHARING:
Plan to Share IPD: No
This item has not yet been defined.

REFERENCES:
- [Background] Hu B, Huang S, Yin L. The cytokine storm and COVID-19. J Med Virol. 2021 Jan;93(1):250-256. doi: 10.1002/jmv.26232. Epub 2020 Sep 30. PMID 32592501
- [Background] Bhaskar S, Sinha A, Banach M, Mittoo S, Weissert R, Kass JS, Rajagopal S, Pai AR, Kutty S. Cytokine Storm in COVID-19-Immunopathological Mechanisms, Clinical Considerations, and Therapeutic Approaches: The REPROGRAM Consortium Position Paper. Front Immunol. 2020 Jul 10;11:1648. doi: 10.3389/fimmu.2020.01648. eCollection 2020. PMID 32754159
- [Background] Sharma BB, Singh S, Sharma VK, Choudhary M, Singh V, Lane S, Lepping P, Krishna M, Copeland J. Psychiatric morbidity in chronic respiratory disorders in an Indian service using GMHAT/PC. Gen Hosp Psychiatry. 2013 Jan-Feb;35(1):39-44. doi: 10.1016/j.genhosppsych.2012.09.009. Epub 2012 Oct 31. PMID 23122486
- [Background] Ryerson CJ, Arean PA, Berkeley J, Carrieri-Kohlman VL, Pantilat SZ, Landefeld CS, Collard HR. Depression is a common and chronic comorbidity in patients with interstitial lung disease. Respirology. 2012 Apr;17(3):525-32. doi: 10.1111/j.1440-1843.2011.02122.x. PMID 22221976
- [Background] Shigemura J, Ursano RJ, Morganstein JC, Kurosawa M, Benedek DM. Public responses to the novel 2019 coronavirus (2019-nCoV) in Japan: Mental health consequences and target populations. Psychiatry Clin Neurosci. 2020 Apr;74(4):281-282. doi: 10.1111/pcn.12988. Epub 2020 Feb 23. No abstract available. PMID 32034840
- [Background] Brooks SK, Webster RK, Smith LE, Woodland L, Wessely S, Greenberg N, Rubin GJ. The psychological impact of quarantine and how to reduce it: rapid review of the evidence. Lancet. 2020 Mar 14;395(10227):912-920. doi: 10.1016/S0140-6736(20)30460-8. Epub 2020 Feb 26. PMID 32112714
- See also: Secretaria de la Salud. Lineamientos De Respuesta Y De Acción En Salud Mental Y Adicciones Para El Apoyo Psicosocial Durante La Pandemia Por Covid-19 En Méxic — https://www.gob.mx/salud/documentos/lineamientos-y-documentos-de-apoyo-en-salud-mental-y-adicciones-ante-el-covid-19